CLINICAL TRIAL: NCT04823234
Title: Lung Ultrasound Signs and Patterns in COVID-19 Pregnant Women - "The PINK-CO Protocol"
Brief Title: Lung Ultrasound Signs and Patterns in COVID-19 Pregnant Women
Acronym: PINK-CO
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Luigi Vetrugno, Clinical Professor in Anesthesiology and Intensive Care, Azienda Sanitaria-Universitaria Integrata di Udine
Other Study IDs: CEUR-2021-223
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Pregnancy Complications; Covid19
MeSH Terms: conditions — Pregnancy Complications; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Lung ultrasound signs in Covid 19 positive pregnant patients

SUMMARY:
SARS-CoV-2 impact on pregnant women is not well known yet. Some authors demonstrated that lung ultrasound can give similar results if compared to chest computed tomography and better results if compared to chest x-rays without radiations and limited risks for mother and fetus.

The Lung Ultrasound Score (LUS) can be used to asses the entity and monitor the evolution of lung impairment.

Some authors described an artifact, the "light beam", as a typical ultrasound sign in COVID-19 positive patients.

With our study we hypothesize to understand the prevalence of this sign and other ultrasound signs in pregnant COVID-19 positive patients.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant COVID 19 positive patients admitted at our institution who had lung ultrasound performed

Exclusion Criteria:

* are < 18 years old
* history of rheumatic disease
* history of spontaneous pneumothorax
* fibrothorax
* history of thoracic surgery
* no consent given

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All pregnant COVID 19 positive patients admitted at our institution
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Light Beam | 24 hours after admission
  Evaluate the prevalence of the light beam sign

SECONDARY OUTCOMES:
Ultrasound patterns | 24 hours after admission
  Evaluate the prevalence of ultrasound signs and patterns during pregnancy
Lung ultrasound score | 24 hours after admission
  Evaluate if the Lung ultrasound score relates with the clinical presentation of the patient
Illness severity | 24 hours after admission
  Evaluate if the lung ultrasound score relates with the prognosis
Length of stay | 24 hours after admission
  Evaluate if the lung ultrasound score relates with the length of stay

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Intensive Care Clinic - Department of Medicine - ASUIUD, Udine, Italy

REFERENCES:
- [Background] Rasmussen SA, Smulian JC, Lednicky JA, Wen TS, Jamieson DJ. Coronavirus Disease 2019 (COVID-19) and pregnancy: what obstetricians need to know. Am J Obstet Gynecol. 2020 May;222(5):415-426. doi: 10.1016/j.ajog.2020.02.017. Epub 2020 Feb 24. PMID 32105680
- [Background] Li J, Long X, Wang X, Fang F, Lv X, Zhang D, Sun Y, Hu S, Lin Z, Xiong N. Radiology indispensable for tracking COVID-19. Diagn Interv Imaging. 2021 Feb;102(2):69-75. doi: 10.1016/j.diii.2020.11.008. Epub 2020 Nov 24. PMID 33281082
- [Background] Vetrugno L, Bove T, Orso D, Barbariol F, Bassi F, Boero E, Ferrari G, Kong R. Our Italian experience using lung ultrasound for identification, grading and serial follow-up of severity of lung involvement for management of patients with COVID-19. Echocardiography. 2020 Apr;37(4):625-627. doi: 10.1111/echo.14664. Epub 2020 Apr 15. PMID 32239532
- [Background] Convissar DL, Gibson LE, Berra L, Bittner EA, Chang MG. Application of Lung Ultrasound During the COVID-19 Pandemic: A Narrative Review. Anesth Analg. 2020 Aug;131(2):345-350. doi: 10.1213/ANE.0000000000004929. PMID 32366774
- [Background] Lichtenstein D. Lung ultrasound in the critically ill. Curr Opin Crit Care. 2014 Jun;20(3):315-22. doi: 10.1097/MCC.0000000000000096. PMID 24758984
- [Background] Bouhemad B, Mongodi S, Via G, Rouquette I. Ultrasound for "lung monitoring" of ventilated patients. Anesthesiology. 2015 Feb;122(2):437-47. doi: 10.1097/ALN.0000000000000558. No abstract available. PMID 25501898
- [Background] Lichter Y, Topilsky Y, Taieb P, Banai A, Hochstadt A, Merdler I, Gal Oz A, Vine J, Goren O, Cohen B, Sapir O, Granot Y, Mann T, Friedman S, Angel Y, Adi N, Laufer-Perl M, Ingbir M, Arbel Y, Matot I, Szekely Y. Lung ultrasound predicts clinical course and outcomes in COVID-19 patients. Intensive Care Med. 2020 Oct;46(10):1873-1883. doi: 10.1007/s00134-020-06212-1. Epub 2020 Aug 28. PMID 32860069
- [Derived] Vetrugno L, Sala A, Orso D, Meroi F, Fabbro S, Boero E, Valent F, Cammarota G, Restaino S, Vizzielli G, Girometti R, Merelli M, Tascini C, Bove T, Driul L; PINK-CO study investigators. Lung Ultrasound Signs and Their Correlation With Clinical Symptoms in COVID-19 Pregnant Women: The "PINK-CO" Observational Study. Front Med (Lausanne). 2022 Jan 21;8:768261. doi: 10.3389/fmed.2021.768261. eCollection 2021. PMID 35127744